CLINICAL TRIAL: NCT05986877
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending-Dose Phase Ia Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of STSA-1201 Injection in Healthy Subjects
Brief Title: A Study of STSA-1201 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Staidson (Beijing) Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STSA-1201-01
Record Dates: First submitted 2023-08-03; First posted 2023-08-14 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- lowest dose group (Experimental): 8 subjects will be randomized to receive lowest dose of STSA-1201 or dose-matched placebo.
  Interventions: Drug: STSA-1201 Subcutaneous injection; Drug: Placebo
- low dose group (Experimental): 12 subjects will be randomized to receive low dose of STSA-1201 or dose-matched placebo.
  Interventions: Drug: STSA-1201 Subcutaneous injection; Drug: Placebo
- middle dose group (Experimental): 12 subjects will be randomized to receive middle dose of STSA-1201 or dose-matched placebo.
  Interventions: Drug: STSA-1201 Subcutaneous injection; Drug: Placebo
- high dose group (Experimental): 12 subjects will be randomized to receive high dose of STSA-1201 or dose-matched placebo.
  Interventions: Drug: STSA-1201 Subcutaneous injection; Drug: Placebo

INTERVENTIONS:
Drug: STSA-1201 Subcutaneous injection — Subcutaneous injection
Drug: Placebo — Subcutaneous injection

SUMMARY:
This study is a Phase Ia, randomized, double-blind, placebo-controlled, single dose, dose escalation safety, tolerability, and pharmacokinetic study of STSA-1201 injection in healthy subjects. A total of 44 healthy subjects were enrolled in four dosage groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects, male or female, aged between 18 and 50 years, inclusive.
* Male subjects must have a weight range of 50.0 kg to 75.0 kg inclusive, and female subjects must have a weight range of 45.0 kg to 75.0 kg inclusive. All subjects must have a body mass index (BMI) of 19.0 to 26.0 kg/m^2 inclusive.
* Subjects (and their partners) must abstain from sperm/egg donation and commit to using effective methods of birth control during the trial and for 6 months post-trial.
* Subjects must have a normal or clinically acceptable medical history, physical examination, laboratory test results, chest X-ray and electrocardiogram (ECG).
* Subjects must fully understand the trial procedures, potential adverse reactions, and sign the informed consent form (ICF).

Exclusion Criteria:

* Subjects with significant clinical disorders or conditions (including but not limited to gastrointestinal, rental, liver, neurological, hematologic, endocrine, oncologic, pulmonary, immunologic, psychiatric, or cardiovascular diseases) and subjects with active or suspected infections (viral, fungal, or parasitic).
* Subjects who underwent major surgery within 2 months prior to screening.
* Subjects with allergic constitution (such as allergies to two or more drugs, foods, and pollen) or potential allergy to the trial product/components.
* Subjects positive for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), human immunodeficiency virus antibody (HIV Ab) or treponema pallidum antibody (TP Ab).
* Subjects with Ig E levels exceeding the normal upper limit.
* Subjects who have smoked more than an average of 5 cigarettes per day within the 3 months prior to screening, or who are unable to abstain from using any tobacco or nicotine-containing products during the trial.
* Subjects with a history of alcohol abuse (more than 14 units per week: 1 unit of alcohol =360mL beer or 45mL spirits with 40% alcohol or 100mL wine) within the 6 months prior to screening, or unable to abstain during the trial, or failed alcohol breath test.
* Subjects with drug abuse history (morphine, ketamine, THC, methamphetamine, methylene-dioxymethamphetamine, cocaine) within 1 year prior to screening or those testing positive for urine drug abuse screening.
* Subjects who donated or lost > 400 mL blood within 3 months prior to screening, received blood transfusions or products within 4 weeks prior to enrollment, or plan to donate blood during the trial and 3 months post-trial.
* Subjects who participated in another clinical trial or received investigational drugs/vaccines within 3 months prior to screening.
* Subjects who received biologicals or monoclonal antibodies within 3 months prior to screening; subjects who used any medication (including prescription medications, over the counter medications and herbal medicines) within 14 days prior to screening; subjects previously treated with any drugs targeting thymic stromal lymphopoietin (TSLP).
* Subjects consuming xanthine-rich foods/beverages (such as coffee, strong tea, chocolate) or those that affect drug absorption, distribution, metabolism, and excretion within 48 hours prior to administration.
* Subjects who used long-acting estrogen or progestogen injections or implants within 6 months prior to screening or short-acting contraceptives within 30 days prior to the trial.
* Female subjects who test positive for serum human chorionic gonadotropin (HCG) or have abnormal HCG levels exceeding the normal upper limit.
* Female subjects who are pregnant or lactating.
* Subjects with venipuncture intolerance, history of transfusion issues, or blood/ needle-phobia.
* Subjects with any condition or circumstance which, in the opinion of the Investigator, may compromise the ability to provide informed consent, comply with the study protocol, potentially influence study outcomes, jeopardize their own safety, or any other situation deemed unsuitable for study participation by the investigator.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-08-04 (Actual); Primary Completion 2024-03-14 (Actual); Study Completion 2024-03-14 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Clinically Significant Laboratory Abnormalities, Clinically Significant Electrocardiogram、Vital Signs And Physical Examination Abnormalities. | Day0 through Day84
  To evaluate the safety and tolerability of single subcutaneous administration of STSA-1201 in healthy adult subjects.

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Area under the plasma concentration-time curve over a dosing interval, from time 0 to time t (AUC0-t). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Area under the plasma concentration-time curve from time 0 to infinity (AUC0-∞). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Time of maximum concentration (Tmax). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Elimination half-life (t1/2). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Apparent clearance (CL/F). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Apparent volume of distribution (Vz/F). | Day0 through Day84
  To evaluate the single dose pharmacokinetics (PK) characteristics of STSA-1201 in healthy adult subjects.
Change from baseline in concentration of anti-drug antibody. | Day0 through Day84
  To evaluate the immunogenicity of STSA-1201 in healthy subjects:

CONTACTS AND LOCATIONS:
Overall Officials: Xinghe Wang, MD, Principal Investigator — Beijing Shijitan Hospital, Capital Medical University
Locations (1):
- Beijing Shijitan Hospital, Capital Medical University, Beijing, Beijing Municipality, China